CLINICAL TRIAL: NCT01410786
Title: A Comparison of Signature Guides and Conventional Instrumentation With the Oxford Partial Knee System Pilot Study
Brief Title: Oxford Partial Knee Comparative Instrument Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ORTHO.CR.GK1 (407)
Record Dates: First submitted 2011-07-14; First posted 2011-08-05 (Estimated); Last update posted 2017-08-02 (Actual); Status verified 2017-08

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional Oxford instrumentation (Active Comparator): Patients who receive an Oxford Partial Knee with Conventional instrumentation.
  Interventions: Procedure: Conventional Instrumentation
- Signature Guides Oxford (Experimental): Patients who receive an Oxford Partial Knee with Signature Custom Guides
  Interventions: Procedure: Signature Custom Guides

INTERVENTIONS:
Procedure: Conventional Instrumentation — Standard Oxford surgical instruments
  Arms: Conventional Oxford instrumentation
Procedure: Signature Custom Guides — Signature Custom Guides used with Instruments in surgical technique
  Arms: Signature Guides Oxford

SUMMARY:
The purpose of this prospective clinical data-collection is to document the performance and clinical outcomes of the Oxford Partial Knee System using Signature Custom Guides and Conventional Instrumentation.

DETAILED DESCRIPTION:
The purpose of this prospective clinical data-collection is to document the performance and clinical outcomes of the Oxford Partial Knee System using Signature Custom Guides and Conventional Instrumentation.

The FDA has approved the Oxford Partial Knee via Premarket Approval P010014. Also, by being CE marked, the Oxford Partial Knee also conforms to the essential requirements of EC Directive 93/42/EEC; in accordance to 13485:2003. The data gathered will be collated and used to provide feedback to design engineers, support marketing efforts, answer potential questions from reimbursement agencies, and will serve as a part of Biomet's Post Market Surveillance System.

Surgical techniques and patient care are to be standard for the surgeon participating in the protocol for both treatment groups and should be maintained the same throughout the course of the data-collection. There will be no experimental or investigational devices used. There will be no experimental or investigational surgical techniques used. The devices and products will be used in accordance with their instructions for use and/or approved labeling. Any use of the device or collection of clinical data outside of the United States should comply with all local, state, and/or national and international regulations.

ELIGIBILITY:
Inclusion Criteria:

Outside the United States:

-The Oxford Partial Knee System is intended for use in individuals with osteoarthritis or avascular necrosis limited to the medial compartment of the knee and is intended to be implanted with bone cement (in the United States). Use of cementless femoral fixation is permitted outside of the United States only (if it complies with all local, state, and/or national and international regulations), however the same technique must be used consistently throughout the course of the study (cemented or cementless).

Exclusion Criteria:

* The exclusion criteria will include the same contraindications stated in the FDA approved labeling for the device (approved in PMA P010014). These contraindications include:
* Infection, sepsis, and osteomyelitis
* Use in the lateral compartment of the knee
* Rheumatoid arthritis or other forms of inflammatory joint disease
* Revision of a failed prosthesis, failed upper tibial osteotomy or post-traumatic arthritis after tibial plateau fracture
* Insufficiency of the collateral, anterior, or posterior cruciate ligaments which would preclude stability of the device
* Disease or damage to the lateral compartment of the knee
* Uncooperative patient or patient with neurologic disorders who is incapable of following directions
* Osteoporosis
* Metabolic disorders which may impair bone formation
* Osteomalacia
* Distant foci of infections which may spread to the implant site
* Rapid joint destruction, marked bone loss, or bone resorption apparent on roentgenogram
* Vascular insufficiency, muscular atrophy, neuromuscular disease
* Incomplete or deficient soft tissue surrounding the knee
* Charcot's disease
* A fixed varus deformity (not passively correctable) of greater than 15 degrees
* A flexion deformity greater than 15 degrees

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2013-06; Primary Completion 2015-05 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Oxford Knee Score | Two Years
  The Oxford Knee Score is a patient administered questionnaire about how they are functioning and feel about their knee.

SECONDARY OUTCOMES:
Average Operative Time | 1 Year
  From incision to incision closure.

CONTACTS AND LOCATIONS:
Overall Officials: Rod Maxwell, Principal Investigator — Canterbury Orthopaedic Services
Locations (1):
- Leinster Orthopaedic Centre, Christchurch, New Zealand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Insall JN, Dorr LD, Scott RD, Scott WN. Rationale of the Knee Society clinical rating system. Clin Orthop Relat Res. 1989 Nov;(248):13-4. PMID 2805470
- [Background] Dawson J, Fitzpatrick R, Murray D, Carr A. Questionnaire on the perceptions of patients about total knee replacement. J Bone Joint Surg Br. 1998 Jan;80(1):63-9. doi: 10.1302/0301-620x.80b1.7859. PMID 9460955